CLINICAL TRIAL: NCT06614725
Title: A Phase 3, Randomized, Placebo-controlled, Observer-blind Study in India to Evaluate Immune Response, Reactogenicity and Safety of a Single Intramuscular Dose of RSVPreF3 OA Investigational Vaccine When Administered to Older Adults >=60 Years of Age and Adults 50-59 Years of Age at Increased Risk of Respiratory Syncytial Virus Lower Respiratory Tract Disease
Brief Title: A Study in India on the Immune Response and Safety of a Respiratory Syncytial Virus (RSV) Older Adults (OA) Vaccine When Given to Older Adults 60 Years of Age and Above and Adults 50-59 Years of Age at Increased Risk (AIR) of Respiratory Syncytial Virus Lower Respiratory Tract Disease (RSV-LRTD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 221265
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; Respiratory Syncytial Virus; RSVPreF3 OA vaccine; Immunogenicity; Safety; Reactogenicity; At increased risk (AIR); Older Adults; Respiratory syncytial virus lower respiratory tract disease (RSV-LRTD)
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- OA-RSV group (Experimental): Older adult (OA) participants, greater than or equal to (≥) 60 years of age (YOA), received a single dose of RSVPreF3 OA investigational vaccine at Day 1.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- OA-Placebo group (Placebo Comparator): OA participants, ≥ 60 YOA, received a single dose of placebo at Day 1.
  Interventions: Combination Product: Placebo
- Adults-AIR-RSV group (Experimental): Adult participants, 50-59 YOA, at increased risk (AIR) of Respiratory Syncytial Virus - Lower Respiratory Tract Disease (RSV-LRTD), received a single dose of RSVPreF3 OA investigational vaccine at Day 1.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- Adults-AIR-Placebo group (Placebo Comparator): Adult participants, 50-59 YOA, at increased risk (AIR) of RSV-LRTD, received a single dose of placebo at Day 1.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — 1 dose of RSVPreF3 OA investigational vaccine administered intramuscularly on Day 1 to participants in OA-RSV and Adults-AIR-RSV groups.
  Arms: Adults-AIR-RSV group; OA-RSV group
Combination Product: Placebo — 1 dose of placebo (saline solution) administered intramuscularly on Day 1 to participants in OA-Placebo and Adults-AIR-Placebo groups.
  Arms: Adults-AIR-Placebo group; OA-Placebo group

SUMMARY:
The purpose of the study is to evaluate the immunogenicity and safety of a single dose of investigational RSVPreF3 OA vaccine in Indian older adults 60 years of age (YOA) and above and Indian adults 50-59 YOA at increased risk of RSV-LRTD.

ELIGIBILITY:
Inclusion Criteria:

Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol.

• Written or witnessed informed consent obtained from the participant (participant must be able to understand the informed consent) prior to performance of any study-specific procedure.

Specific inclusion criteria for all participants in Cohort 1 (Older adults)

* Male or female, >= 60 YOA at the time of the study intervention administration.
* Participants who are medically stable in the opinion of the investigator at the time of study intervention administration. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes mellitus, hypertension, or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.
* Participants living in the general community or in an assisted-living facility that provides minimal assistance can be enrolled, such that the participant is primarily responsible for self-care and activities of daily living.

Specific inclusion criteria for all participants in Cohort 2 (Adults-AIR)

* Male or female, 50-59 YOA at the time of the study intervention administration.
* Participants should be diagnosed with at least 1 of the following medical conditions and considered medically stable by the investigator:
* Chronic pulmonary disease resulting in activity restricting symptoms or use of long term medication:

  * Chronic obstructive pulmonary disease (COPD)
  * Asthma
  * Cystic fibrosis
  * Other chronic respiratory diseases: lung fibrosis, restrictive lung disease, interstitial lung disease, emphysema, or bronchiectasis
* Chronic cardiovascular disease:

  * Chronic heart failure (CHF)
  * Pre-existing coronary artery disease (CAD not otherwise specified)
  * Cardiac arrhythmia
* Diabetes mellitus: type 1 or type 2

Other diseases at increased risk for RSV-LRTD disease:

* Chronic kidney disease
* Chronic liver disease

  * Female participants of non-childbearing potential may be enrolled in the study. Non childbearing potential is defined as hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or post-menopause.
  * Female participants of childbearing potential may be enrolled in the study if the participant
* has practiced adequate contraception from 1 month prior to study intervention administration, and
* has a negative pregnancy test on the day of and prior to study intervention administration, and
* has agreed to continue adequate contraception for at least 1 month after the study intervention administration.

Exclusion Criteria:

Medical Conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, resulting from disease (e.g. current malignancy, human immunodeficiency virus) or immunosuppressive/cytotoxic therapy (e.g., medication used during cancer chemotherapy, organ transplantation, or to treat autoimmune disorders), based on medical history and physical examination (no laboratory testing required).
* Unstable chronic illness.
* Recurrent history or uncontrolled neurological disorders or seizures. Participants with medically-controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol (e.g. completion of the eDiary, attend phone call/study site visits).
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study (e.g., life-threatening disease).
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant Therapy

* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study interventions during the period beginning 30 days (Day -29 to Day 1) before the dose of study interventions or their planned use during the study period (Day 1 up to Month 6).
* Previous vaccination with licensed or investigational RSV vaccine. Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the dose of study intervention administration, with the exception of inactivated, subunit and split influenza vaccines or COVID-19 vaccines (fully licensed or with emergency use authorization [EUA]) which can be administered up to 14 days before or from 14 days after the study intervention administration.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

  * Up to 3 months prior to the study intervention administration:
  * For corticosteroids, this will mean prednisone equivalent >= 20 mg/day for adult participants. Inhaled and topical steroids are allowed.
  * Administration of immunoglobulins and/or any blood products or plasma derivatives.
  * Up to 6 months prior to study intervention administration: long-acting immune modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies, antitumoral medication.

Prior/Concurrent Clinical Study Experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other Exclusion Criteria for all participants

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Participation of any study personnel or their immediate dependents, family, or household members.
* Planned move during the study conduct that prohibits participation until study end.
* Bedridden participants.

Other Exclusion Criteria for cohort 2 (Adults-AIR)

* Pregnant or lactating female participant.
* Female participant planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
RSV-A neutralizing titers expressed as Geometric Mean Titers (GMTs) | At Day 1 (pre-study intervention administration)
  RSV-A neutralizing titers are given as GMTs and are expressed as Estimated Dilution 60 (ED60).
RSV-A neutralizing titers expressed as GMTs | At Day 31 (1 month post-study intervention administration)
  RSV-A neutralizing titers are given as GMTs and are expressed as ED60.
RSV-B neutralizing titers expressed as GMTs | At Day 1 (pre-study intervention administration)
  RSV-B neutralizing titers are given as GMTs and are expressed as ED60.
RSV-B neutralizing titers expressed as GMTs | At Day 31 (1 month post-study intervention administration)
  RSV-B neutralizing titers are given as GMTs and are expressed as ED60.

SECONDARY OUTCOMES:
Number of participants reporting any solicited administration site events | Day 1 (day of administration) to Day 4
  Assessed solicited administration site adverse events (AEs) were redness (erythema), pain and swelling at administration site. Any = occurrence of the AE regardless of intensity grade or relationship to the study interventions.
Number of participants reporting any solicited systemic events | Day 1 (day of administration) to Day 4
  Assessed solicited systemic events were arthralgia (joint pain), fatigue (tiredness), fever (pyrexia), headache, and myalgia (muscle pain). Fever was defined as temperature ≥38.0 degrees Celsius (°C), regardless of the location of measurement. The route for measuring temperature could be oral or axillary. Any = occurrence of the symptom regardless of intensity grade or relationship to the study interventions.
Number of participants reporting any unsolicited AEs | Day 1 to Day 30
  An unsolicited AE was an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs included both serious and non-serious AEs, and potential immune-mediated diseases (pIMDs). Any = occurrence of the event regardless of intensity grade or relation to the study intervention.
Number of participants reporting any serious adverse events (SAEs) | From Day 1 up to data lock point of primary analysis (median follow-up: 176 days)
  An SAE was any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, is considered or defined as an important medical event, or abnormal pregnancy outcomes. Any = occurrence of the event regardless of the intensity grade or relation to the study intervention.
Number of participants reporting any SAEs | From Day 1 up to study end (approximately 6 months post study intervention administration)
  Data not available at the time of initial results posting will be updated at the final results disclosure stage.
Number of participants reporting any pIMDs | From Day 1 up to data lock point of primary analysis (median follow-up: 176 days)
  pIMDs were a subset of adverse events of special interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. Any = occurrence of the event regardless of the intensity grade or relation to the study intervention.
Number of participants reporting any pIMDs | From Day 1 up to study end (approximately 6 months post study intervention administration)
  Data not available at the time of initial results posting, will be updated at the final results disclosure stage.

CONTACTS AND LOCATIONS:
Locations (13):
- India (13):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Aligarh
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Darjeeling
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Kanpur
  - GSK Investigational Site, Kelambākkam
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Pune-411 043
  - GSK Investigational Site, Raipur
  - GSK Investigational Site, Vadu Budruk Pune

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/